CLINICAL TRIAL: NCT03995940
Title: Neurological Outcomes of Primary Intracerebral Haemorrhage Admitted in Intensive Care Unit at the University Hospital of Grenoble Alpes
Brief Title: Neurological Outcomes of Primary Intracerebral Haemorrhage
Acronym: HIP-REA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.029; 2019-A00345-52 (Other: ID RCB)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Intracranial Hemorrhage, Hypertensive
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to determine the one-year neurological outcome of patients admitted to an intensive care unit (ICU) for a primary and spontaneous supratentorial intracerebral hemorrhages (ICH).

DETAILED DESCRIPTION:
ICH represent a diagnostic and therapeutic emergency. ICH account for 20% of strokes with a one-year mortality of more than 45% and an uncertain neurological outcome.

For ICH patients, the main initial challenge is to determine the long term neurological outcomes and adapt the therapeutic strategy.

The majority of primary and spontaneous ICH studies involve patients in stroke units.

The study is an observational type 3 research with all the patients admitted in all the University Hospital of Grenoble Alpes ICUs between July 2012 and July 2017 for a primary and spontaneous supratentorial ICH

ELIGIBILITY:
Inclusion Criteria:

* Admission in one of the four University Hospital of Grenoble Alpes ICUs between July 2012 and July 2017 for primary and spontaneous supratentorial ICH.
* Not opposed to participate in a research protocol (asked by phone call)

Exclusion Criteria:

* Pediatric patient
* Infra-tentorials ICH
* No spontaneous ICH (after head trauma)
* Secondary ICH (anevrisum, arteriovenous malformation, tumor, hemorrhagic transformation, vascularitis)
* Persons referred to in Articles L1121-5 to L1121-8 of the french public health code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a primary and spontaneous supratentorial ICH
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Neurological outcomes | One year after the stroke
  Collection of the Modified Ranking Scale (mRS) at one year by patients phone call or with the medicale file.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided